CLINICAL TRIAL: NCT02783716
Title: Vascular Endothelial Function and Cardiac Resynchronization Response in Patients With Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID and staffing issues study was terminated
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hon-Chi Lee, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-006402
Record Dates: First submitted 2016-05-20; First posted 2016-05-26 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Resynchronization Therapy (CRT) Group (Active Comparator): Participants undergoing Cardiac Resynchronization Therapy Implantation (CRT) implantation for heart failure as part of standard of care will receive EndoPAT testing and collection of subcutaneous adipose tissue
  Interventions: Procedure: Subcutaneous adipose tissue collection; Diagnostic Test: Peripheral arterial tonometry (PAT)
- Control Group (Active Comparator): Participants undergoing device pacemaker or implantable cardioverter-defibrillator (ICD) implantation or pack change for sinus node dysfunction or Atrioventricular (AV) block as part of standard of care will receive EndoPAT testing and collection of subcutaneous adipose tissue
  Interventions: Procedure: Subcutaneous adipose tissue collection; Diagnostic Test: Peripheral arterial tonometry (PAT)

INTERVENTIONS:
Procedure: Subcutaneous adipose tissue collection — During standard of care device implantation procedure, a small piece of fat tissue will be removed from the device pocket inside the chest
Diagnostic Test: Peripheral arterial tonometry (PAT) — Non-invasive testing for blood vessel function. Specially designed finger probes placed on the middle finger of each hand. Pulsatile volume changes of the distal digit inducing pressure alterations in the finger cuff will be sensed by pressure transducers and recorded. Endothelial function will be measured via a reactive hyperemia (RH)-PAT index (RHI)
  Other Names: EndoPAT

SUMMARY:
The purpose of this research study is to determine the role of blood vessel endothelial function in heart failure and the effect of Cardiac Resynchronization Therapy (CRT) on heart and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* CRT Group: Patients recommended for CRT-P or CRT-D for heart failure (HF) according to current American Heart Association (AHA)/American College of Cardiology (ACC)/Heart Rhythm Society (HRS) guidelines of Left Ventricle Ejection Fraction (LVEF)<35%, Left Bundle Branch Block (LBBB)>120 ms, New York Heart Association (NYHA) Class II-III).
* Control Group: Patients who undergo device (pacemaker or ICD) implantation or a pack change for sinus node dysfunction or AV blocks

Exclusion Criteria:

* Patients who are unwilling or unable to return for follow up visits 3 months after device implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05; Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function | baseline, 3 months
  Vascular endothelial function will be measured using peripheral arterial tonometry as the reactive hyperemia index (RHI) at baseline and at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Chi Lee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials